CLINICAL TRIAL: NCT01387919
Title: Time Course and Nature of Nutrient Sensing During Fasting in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Centre for Medical Systems Biology (Unknown)
Responsible Party: Hanno Pijl, Leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P10.164
Record Dates: First submitted 2011-07-01; First posted 2011-07-06 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-01

CONDITIONS: Nutrient Sensing During a Prolonged Fast
Keywords: Set time points during 48 hours of fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): healthy young and lean men
  Interventions: Behavioral: Prolonged fasting

INTERVENTIONS:
Behavioral: Prolonged fasting — 48 hours of fasting

SUMMARY:
Several studies have begun to determine the time course of events sensing energy availability in rodents. In contrast, there is not a single study that has examined this in humans to date. A better understanding of this energy sensing machinery in humans is of utmost importance to give us new insights into developing new therapies for common diseases such as obesity, diabetes mellitus, cardiovascular diseases and cancer. In these diseases, disturbances in the energy-sensing machinery possibly play a role. To determine the time course of energy sensing events in humans, the investigators will measure the concentration of various hormones in plasma, and biochemical changes in skeletal muscle at sequential time points during starvation in humans. The investigators choose to study the molecular machinery in muscle, since muscle is very sensitive to fuel deprivation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age 19-29 years old
* Body mass index (BMI) 19-25 kg/m2
* Stable weight for the last 3 months
* Caucasian
* Fasting plasma glucose (FPG) < 6 mmol/L
* Well-controlled blood pressure (< 150/95 mmHg)
* Creatinine <100 umol/l
* Hb > 7.5 mmol/l
* Negative family history (first degree) of type 2 diabetes mellitus (DM2)

Exclusion Criteria:

* Use of medication known to affect glucose metabolism (for example prednisone) or lipid metabolism
* Significant (chronic) disease
* Smoking (current)
* Alcohol consumption of more than 14 units per week at present or in the past
* Difficult accessible veins for insertion of an intravenous catheter
* Recent blood donation (within the last 3 months)
* Recent participation in other research projects (within the last 3 months), participation in 2 or more projects in one year
* Rigorous exercise/sports 5 or more days a week

Ages: 19 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in several proteins/ribonucleic acid (RNA) from muscle biopsies upon fasting | 1.5h, 4h, 10h, 24h

SECONDARY OUTCOMES:
Change in several hormones, lipids etc. from blood samples upon fasting | 1.5h, 4h, 10h, 24h

CONTACTS AND LOCATIONS:
Overall Officials: Hanno Pijl, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands